CLINICAL TRIAL: NCT04065490
Title: A Double-Masked, Randomized, Sham-Controlled, Parallel Group, Multi-Center Study to Assess the Safety and Efficacy of Photobiomodulation (PBM) in Subjects With Dry Age-Related Macular Degeneration (AMD) (LIGHTSITE III)
Brief Title: Study of Photobiomodulation to Treat Dry Age-Related Macular Degeneration (LIGHTSITE III)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: LumiThera, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CSP005
Record Dates: First submitted 2019-08-16; First posted 2019-08-22 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2021-02

CONDITIONS: Dry Age-related Macular Degeneration
Keywords: Dry age-related macular degeneration; Photobiomodulation; Visual Acuity; Contrast Sensitivity; Drusen; Optical coherence tomography

STUDY DESIGN:
Intervention Model Description: Valeda Light Delivery System
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- PBM Treatment (Experimental): The Valeda™ Light Delivery System
  Interventions: Device: Valeda PBM treatment
- Sham Treatment (Sham Comparator): The Valeda™ Light Delivery System non-effective treatment
  Interventions: Device: Valeda Sham treatment

INTERVENTIONS:
Device: Valeda PBM treatment — The Valeda Light Delivery System
  Arms: PBM Treatment
Device: Valeda Sham treatment — The sham mode of the Valeda Light Delivery System.
  Arms: Sham Treatment

SUMMARY:
This LIGHTSITE III study is a double-masked, sham-controlled, parallel design, prospective multi-site study for the use of PBM as a treatment for visual impairment in subjects with dry AMD.

DETAILED DESCRIPTION:
This study is a double-masked, sham-controlled, parallel design prospective, multi-site study on the use of photobiomodulation (PBM) as a treatment for visual impairment in subjects with dry AMD. Subjects will receive repeated sham or PBM treatments at several time-points throughout the 2-year study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female at least 50 years of age at Screening visit
2. ETDRS BCVA letter score of between 50* and 75* (Snellen equivalent of 20/100 to 20/32). *If the subject meets this criterion at the Screening Visit, but the Baseline BCVA letter score is between 48 and 77, the subject may be entered in the study.
3. Diagnosis of dry AMD as defined by the presence of the following:

   Drusen that are intermediate in size or larger (63 μm or larger in diameter) with at least a few (3) being regular drusen and not pseudodrusen and/or geographic atrophy (GA) visible on two of the following: color fundus images, OCT and/or FAF, to be confirmed by the reading center
4. Able to communicate well with the Investigator and able to understand and comply with the requirements of the study
5. Informed of the nature of this study and has provided written, informed consent in accordance with institutional, local and national regulatory guidelines

Exclusion Criteria:

1. Current or history of neovascular maculopathy that includes any of the following (to be confirmed by the reading center):

   1. Choroidal neovascularization (CNV) defined as pathologic angiogenesis originating from the choroidal vasculature that extends through a defect in Bruch's membrane
   2. Serous and/or hemorrhagic detachment of the neurosensory retina or retinal pigment epithelial (RPE)
   3. Retinal hard exudates (a secondary phenomenon resulting from chronic intravascular leakage)
   4. Subretinal and sub-RPE fibrovascular proliferation
   5. Disciform scar (subretinal fibrosis)
2. Presence of center involving GA within the central ETDRS 1 mm diameter at Screening, to be confirmed by the reading center
3. Media opacities, including cataracts, which might interfere with visual acuity or imaging in the study eye(s). Subjects should not be entered if there is likelihood that they will require cataract surgery in the study eye in the next 24 months.
4. Posterior capsule opacification, which might interfere with visual acuity or imaging in the study eye(s). Subjects should not be entered if there is likelihood that they will require surgery in the study eye in the next 24 months.
5. Invasive eye surgery (e.g. cataract, capsulotomy) on a qualifying eye within three 3 months prior to Screening
6. Ocular disorder or disease that partially or completely obstructs the pupil (e.g. posterior synechia in uveitis)
7. Visually significant disease in any ocular structure apart from dry AMD (e.g. diabetic macular edema, glaucoma (using >2 eye drop medications, uncontrolled IOP and/or central/paracentral visual field loss), glaucoma surgery, active uveitis, active vitreous disease, intraocular tumor, retinal vascular diseases)
8. Ocular disorder or disease other than dry AMD that could cause drusen (glomerulonephritis Type 2, Autosomal dominant drusen), GA (North Carolina dystrophy) or mitochondrial diseases (parafoveal petaloid GA, Stargardt disease)
9. Presence or history of disease or condition affecting functional vision without obvious structural abnormalities (e.g. amblyopia, stroke, nystagmus)
10. Serious medical illness that will prevent the subject from performing study activities (including cardiac, hepatic, renal, respiratory, endocrinologic, neurologic, or hematologic disease) or, in the judgement of the Investigator, is likely to require surgical intervention or hospitalization at any point during the study
11. Presence of or history of malignancy within the past 5 years other than non-melanoma skin or squamous cell cancer or cervical carcinoma in-situ
12. Is non-ambulatory
13. Presence or history of known light sensitivity to yellow light, red light, or near infrared radiation (NIR), or if they have a history of light activated CNS disorders (e.g. epilepsy, migraine)
14. Use of any photosensitizing agent (e.g. topicals, injectables, oral) within 30 days of treatment without consulting subject's physician
15. History of drug, alcohol or substance abuse within 3 months prior to Screening
16. Has received an investigational drug or treatment with an investigational device within 3 months prior to Screening
17. If on any anti-oxidant or vitamin Age-Related Eye Disease Study (AREDS) supplement for dry AMD, has not been stabilized for a minimum of 1 month prior to Screening. Subjects are considered to be stable if they are taking the AREDS supplements consistently as prescribed by their treating doctor.
18. Has received Low Vision Rehab/Therapy within 30 days prior to Screening or intends to receive during the study
19. Has an open sore(s) that may come in contact with the Valeda System, has periorbital skin erythema or is prone to such conditions with exposure to light.
20. In the opinion of the Investigator, is unlikely to comply with the study protocol

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Best Corrected Visual Acuity | 21 months
  Mean change from baseline in BCVA.

SECONDARY OUTCOMES:
Contrast Sensitivity | 21 months
  Mean change from baseline (pre-treatment) in contrast sensitivity at 40 cm.
Central Drusen Volume | 21 Months
  Mean change from baseline (pre-treatment) in central Drusen volume.
Central Drusen Thickness | 21 Months
  Mean change from baseline (pre-treatment) in central Drusen thickness.

OTHER OUTCOMES:
Contrast Sensitivity | 21 Months
  Mean change from baseline (pre-treatment) in contrast sensitivity at 80 cm and 120 cm.
Visual Function Questionnaire | 21 Months
  Mean change from baseline (pre-treatment) in Visual Function Questionnaire (VFQ-25) composite score.
Reading Speed | 21 Months
  Mean change from baseline (pre-treatment) to Month 21 in monocular reading speed assessed by the Radner Reading Chart.
Geographic Atrophy | 21 Months
  Mean change from baseline in the GA lesion area of the PBM treatment group versus the sham treatment group, as measured by FAF.
Low Luminance- Best Corrected Visual Acuity | 21 Months
  Mean change from baseline in the LLBVCA.

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - Retina Vitreous Associates Medical Group, Beverly Hills, California
  - Stanford University, Palo Alto, California
  - Florida Eye Clinic, Altamonte Springs, Florida
  - Cumberland Valley Retina Consultants, Hagerstown, Maryland
  - Mid Atlantic Retina, Cherry Hill, New Jersey
  - New York Ear and Eye Infirmary, New York, New York
  - Duke Eye Center, Durham, North Carolina
  - Cumberland Valley Retina Consultants, Chambersburg, Pennsylvania
  - Gulf Coast Eye Institute, McAllen, Texas
  - Retina Consultants of Houston, The Woodlands, Texas
  - Retina Center Northwest, Silverdale, Washington

IPD SHARING:
Plan to Share IPD: No